CLINICAL TRIAL: NCT00260546
Title: An-Art Study: AV-Node Ablation in Cardiac Resynchronisation Therapy
Brief Title: An-Art Study: Atrioventricular (AV) Node Ablation in Cardiac Resynchronisation Therapy
Status: Withdrawn | Phase: Early Phase 1 | Type: Interventional
Why Stopped: No patients enrolled for 6 months.
Sponsor: University Hospital, Basel, Switzerland (Other)
Responsible Party: Christian Sticherling, MD, University Hospital Basel
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 159/05
Record Dates: First submitted 2005-11-29; First posted 2005-12-01 (Estimated); Last update posted 2011-09-30 (Estimated); Status verified 2011-09

CONDITIONS: Congestive Heart Failure
Keywords: Ventricular dyssynchrony
MeSH Terms: conditions — Heart Failure

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Procedure: AV-node ablation — Patients that are randomized to AV node ablation will have their AV-node ablated using a transfemoral approach. Concurrently,a back-up pacing lead will temporarily be placed in the right ventricle.

SUMMARY:
Cardiac resynchronisation therapy (CRT) is a highly effective treatment option for patients with symptomatic heart failure and electrical intraventricular dyssynchrony, who are unresponsive to medical therapy. CRT has been shown to improve the quality of life in these patients and lately two studies had shown a mortality reduction with and without the adjunct of an implantable cardioverter defibrillator (ICD). Unfortunately, up to 25% of the CRT recipients do not show a symptomatic improvement after device implantation ("non-responder"). Because of possible intermittent tachycardiac intrinsic conduction, it remains difficult in numerous patients to assure a 100% biventricular stimulation as the prerequisite for a beneficial therapeutic effect. In a important study by Knight et al it could be shown that in a population of 440 CRT-patients, 36% did not have continuous biventricular stimulation. The main cause was the occurrence of atrial tachyarrhythmias, in particular atrial fibrillation. The medical control of rapid ventricular conduction remains a difficult problem in heart failure patients. Furthermore it is unknown how many patients have good biventricular pacing under resting conditions but develop an improved AV-conduction with exercise. This can cause inhibition of ventricular stimulation or in many cases fusion beats. Conversely, an AV-interval programmed too short may have detrimental effects on diastolic filling times.

The safest method to control the ventricular rate and prevent ventricular fusion beats with a normal AV time is the AV node ablation using radiofrequency ablation.

The An Art Study investigates whether patients with an implanted CRT pacemaker or a CRT defibrillator will benefit from an AV-node-ablation using a combined symptomatic heart failure endpoint and duration of biventricular stimulation as compared to a CRT control group.

ELIGIBILITY:
Inclusion Criteria:

* All patients who had a CRT pacemaker or CRT-ICD implanted and who are under optimal medical therapy, can be included 3 months after implantation of the device.

Exclusion Criteria:

* The sole exclusion criterion is no consent of the patient.

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2006-05; Primary Completion 2008-12 (Estimated); Study Completion 2008-12 (Estimated)

PRIMARY OUTCOMES:
Percentage of biventricular stimulated heart cycles | 2 years

SECONDARY OUTCOMES:
Combined endpoint of worsening of heart failure, NYHA class, 6-minute walking distance, and hospitalisation for heart failure, death or heart transplantation | 2 years

CONTACTS AND LOCATIONS:
Overall Officials: Christian Sticherling, M.D., Principal Investigator — University Hospital Basel, Cardiology